CLINICAL TRIAL: NCT06049797
Title: A Phase IV, Longitudinal, Observational Study Examining Real-World Outcomes of Non-Hormonal Pharmacotherapies Among Individuals Treated for Bothersome Vasomotor Symptoms
Brief Title: A Study Following Women in Menopause Treated With a Non-hormonal Therapy for Hot Flashes and Night Sweats
Acronym: OPTION-VMS
Status: Active, not recruiting | Type: Observational
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2693-MA-3457
Record Dates: First submitted 2023-09-18; First posted 2023-09-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hot Flashes
Keywords: fezolinetant; vasomotor symptoms; menopause; night sweats; non-hormonal treatment
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant; Paroxetine; Citalopram; Escitalopram; Desvenlafaxine Succinate; Venlafaxine Hydrochloride; Gabapentin; Clonidine; Pregabalin; oxybutynin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neurokinin 3 Receptor (NK3-R) Antagonist: Participants prescribed NK3-R Antagonist for the treatment of VMS.
  Interventions: Drug: Fezolinetant
- Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI): Participants prescribed SSRI/SNRI for the treatment of VMS.
  Interventions: Drug: Paroxetine; Drug: Citalopram; Drug: Escitalopram; Drug: Desvenlafaxine; Drug: Venlafaxine; Drug: Any other SSRI/SNRI not already specified
- Other: Participants prescribed something other than NK3-R Antagonist or SSRI/SNRI for the treatment of VMS.
  Interventions: Drug: Gabapentin; Drug: Clonidine; Drug: Pregabalin; Drug: Oxybutynin; Drug: Any other non-hormonal pharmacologic therapy prescribed for the treatment of VMS not included in a category above

INTERVENTIONS:
Drug: Fezolinetant — Oral
  Other Names: ESN364; VEOZAH
  Groups: Neurokinin 3 Receptor (NK3-R) Antagonist
Drug: Paroxetine — Oral
  Groups: Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI)
Drug: Citalopram — Oral
  Groups: Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI)
Drug: Escitalopram — Oral
  Groups: Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI)
Drug: Desvenlafaxine — Oral
  Groups: Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI)
Drug: Venlafaxine — Oral
  Groups: Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI)
Drug: Gabapentin — Oral
  Groups: Other
Drug: Clonidine — Oral
  Groups: Other
Drug: Pregabalin — Oral
  Groups: Other
Drug: Oxybutynin — Oral
  Groups: Other
Drug: Any other SSRI/SNRI not already specified — Oral
  Groups: Selective serotonin reuptake inhibitor (SSRI)/Serotonin and norepinephrine reuptake inhibitor (SNRI)
Drug: Any other non-hormonal pharmacologic therapy prescribed for the treatment of VMS not included in a category above — Oral
  Groups: Other

SUMMARY:
Hot flashes and night sweats (also known as vasomotor symptoms or VMS) are the most common symptoms which bother women in menopause. This study will follow women going through menopause who have hot flashes and night sweats that cause them bother. They will be starting a non-hormonal therapy prescribed by their healthcare provider (HCP) to treat these symptoms. The women will visit their HCP's office, research center, or both. They will receive prescriptions for the non-hormonal therapy from their HCP for up to 1 year. This real-world study will provide information on outcomes from various non-hormonal therapies. The study sponsor (Astellas) will not decide which therapy the women receive. However, the sponsor will provide instructions on when the women visit their clinic, and what is recorded during the study. Some of the visits will be in-person, but most will be virtual. The virtual visits can be carried out at home using a smartphone, tablet or computer. The main aim of the study is to check if the hot flashes and night sweats that bother women change after 12 weeks (3 months) of treatment. The study will also check the women's sleep patterns, their productivity at work, and their general well-being before and after starting treatment. The overall safety of the non-hormonal therapies will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Participant is diagnosed with bothersome VMS due to/associated with menopause for at least 3 months based on a standard of care assessment captured in consultation with an HCP including the participant's history, routine physical examination, and routine laboratory assessments.
* HCP has made the clinical decision to begin pharmacologic treatment with a non-HT including, a selective neurokinin 3 receptor (NK3-R) antagonist, an SSRI, SNRI, gabapentin, clonidine, pregabalin, oxybutynin or other non-HT, as part of the standard treatment for VMS. This may be the first course of treatment, a restart or a switch from one drug (HT/non- HT) to another non-HT. A restart or switch of a previous therapy requires a minimum of a 10-day period not on therapy/washout period prior to pre-baseline.
* Participant's health status is stable based on their medical history and general physical exam and determined to be a candidate for treatment with non-HTs.
* If participant has been prescribed an SSRI or SNRI for the treatment of depression or anxiety, they must be on a stable or consistent dose for a minimum of 3 months prior to screening.
* Participant has a negative urine pregnancy test at screening if not post-menopausal.
* Only for participants utilizing complementary and alternative therapies, mind-body techniques, or supplements for the treatment of VMS: participant has been on such therapies for ≥ 3 months prior to screening and intends to continue through duration of study.
* Confirmation has been made that the participant is able to obtain the prescribed non hormonal therapy (e.g., insurance coverage verified, participant has ability to self pay, or patient support program activated for at least 12 months for the uninsured participants, if applicable).

Exclusion Criteria:

* Participant is currently enrolled in any interventional or non-interventional wearable device study.
* Participant has any condition which makes the participant unsuitable for the study.
* Participant has a contraindication to the non-HT they are being prescribed for the treatment of VMS.
* Participant is currently taking hormonal contraceptives or other systemic HTs (including estrogen and/or progesterone, and/or testosterone preparations) and has not had a 10-day washout period prior to pre-baseline (vaginal/local estrogen preparations and levonorgestrel-releasing intrauterine system are not prohibited).
* Participant has presence of moderately severe or severe depression per standard of care assessment utilizing a standardized depression screening tool.
* Participant is currently pregnant or planning to become pregnant.
* Participant is post-menopausal and has a history of unexplained uterine bleeding within the last 6 months.
* Participant has pre-existing uncontrolled thyroid disease.
* Participant has unstable angina or participant has uncontrolled hypertension based on a standard of care assessment.

  * Participants who do not meet these criteria may be re-assessed after initiation or review of antihypertensive measures.
  * Participants with a medical history of hypertension can be enrolled once they are medically clear (stable and compliant).
* Participant has had insomnia unrelated to either menopause or bothersome VMS due to/associated with menopause.
* Participant has known substance abuse or alcohol addiction within 6 months of screening.
* Participant has been on intramuscular estradiol within 8 weeks of screening.
* Participant has a current diagnosis of a malignancy or history of a malignancy within the past 2 years (This does not include basal cell carcinoma or breast cancer.)
* Participants with metastatic (Stage 4) breast cancer.
* Participants who have been prescribed adjuvant endocrine therapy (tamoxifen or aromatase inhibitors with or without gonadotropin-releasing hormone analogues) for their non-metastatic (stage 0 to 3) breast cancer but have not maintained a stable treatment regimen for at least 3 months prior to screening.
* Participant has initiated hormone pellet therapy within 6 months of screening.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants experiencing bothersome VMS with a confirmed diagnosis of VMS by an HCP and newly prescribed non-hormonal therapy (non-HT).
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline to week 12 in symptom bother measured by the Menopause-Specific Quality of Life Domain (MENQoL) 1-week recall VMS domain score | Baseline and week 12
  The MENQoL is a 29-item patient reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.

SECONDARY OUTCOMES:
Percentage of participants classified as 1-point responders as measured by the MENQol 1-week recall VMS domain | Up to week 52
  Participants with a reduction (improvement) in symptom bother score ≥ 1 unit will be classified as 1-point responders.
Percentage of participants classified as 2-point responders as measured by the MENQol 1-week recall VMS domain | Up to week 52
  Participants with a reduction (improvement) in symptom bother score ≥ 2 unit will be classified as 2-point responders.
Mean change from baseline in total score of Patient-Reported Outcomes Measurement Information System Sleep Disturbance Sexual Function (PROMIS SD SF) 8b | Baseline and weeks 4, 8, 12, 24 and 52
  The PROMIS SD SF 8b assesses self-reported sleep disturbance over the past 7 days and includes perceptions of restless sleep; satisfaction with sleep; refreshing sleep; difficulties sleeping, getting to sleep or staying asleep; amount of sleep; and sleep quality. Responses to each of the 8 items range from 1 to 5, and the range of possible summed raw scores is 8 to 40. Higher scores on the PROMIS SD SF 8b indicate more of the concept measured (disturbed sleep).
Total score from Patient Global Impression of Severity (PGI-S) of SD | Up to week 52
  The PGI-S SD evaluates patient perceived severity of sleep disturbance. Ratings range from (1) no problems to (4) severe problems.
Total score from Patient Global Impression of Change (PGI-C) of SD | Up to week 52
  PGI-C SD evaluates patient perceived change in sleep disturbance from the initiation of treatment. Ratings range from (1) much better to (7) much worse.
Change from baseline in average daily total sleep time, as recorded by wearable device | Baseline to weeks 4, 8 and 12
  The wearable device will capture movement and physiological signals to derive measures related to sleep.
Change from baseline in average daily sleep efficiency, as recorded by wearable device | Baseline to weeks 4, 8 and 12
  The wearable device will capture movement and physiological signals to derive measures related to sleep.
Change from baseline in average daily wake after sleep onset (WASO), as recorded by wearable device | Baseline to weeks 4, 8 and 12
  The wearable device will capture movement and physiological signals to derive measures related to sleep.
Change from baseline in average daily number of nighttime awakenings, as recorded by wearable device | Baseline to weeks 4, 8 and 12
  The wearable device will capture movement and physiological signals to derive measures related to sleep.
Change from baseline in average daily sleep latency, as recorded by wearable device | Baseline to weeks 4, 8 and 12
  The wearable device will capture movement and physiological signals to derive measures related to sleep.
Mean change from baseline in the MENQoL total score | Baseline to weeks 4, 8, 12, 24 and 52
  The MENQoL is a 29-item patient reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. The total score is the mean of the domain means. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.
Mean change from baseline in the MENQoL vasomotor 1-week recall VMS domain score | Baseline to weeks 4, 8, 24 and 52
  The MENQoL is a 29-item patient reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.
Mean change from baseline in the MENQoL 1-week recall psychosocial domain score | Baseline to weeks 4, 8, 12, 24 and 52
  The MENQoL is a 29-item patient reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.
Mean change from baseline in the MENQoL 1-week recall physical domain score | Baseline to weeks 4, 8, 12, 24 and 52
  The MENQoL is a 29-item patient reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.
Mean change from baseline in the MENQoL 1-week recall sexual domain score | Baseline to weeks 4, 8, 12, 24 and 52
  The MENQoL is a 29-item patient reported outcome (PRO) measure that assesses the impact of 4 domains of menopausal symptoms: vasomotor, psychosocial, physical, and sexual. Each item score ranges from 1 to 8, and each domain is scored separately; each domain mean ranges from 1 to 8. Higher scores represent more bothersome menopausal symptoms. A reduction (improvement) of 1 is the minimum clinically important difference for the MENQoL.
Total score from PGI-C VMS | Up to week 52
  PGI-C VMS evaluates participant perceived change in VMS. Ratings range from (1) much better to (7) much worse.
Mean change from baseline in the VMS-related work productivity and activity impairment (WPAI-VMS) domain score | Baseline to weeks 4, 8, 12, 24 and 52
  The WPAI-VMS is a 6-item PRO measure that examines VMS-related work productivity and activity in the preceding 7 days. It consists of 4 domains: absenteeism, presenteeism, overall work productivity loss, and activity impairment. WPAI-VMS outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity (that is, worse outcomes).
Mean change from baseline in the female sexual function index (FSFI) domain score | Baseline to weeks 4, 8, 12, 24 and 52
  The FSFI is comprised of 19 questions with response options varying among items and ranging from 0 to 5 or 1 to 5. The FSFI has 6 domains: desire, arousal, lubrication, orgasm, satisfaction and pain. Within the individual domains, a domain score of zero indicates that the participant-reported having no sexual activity during the past month. The overall score can range from 2 to 36. A higher score overall or for individual domains indicates better sexual function.
Mean change from baseline in the mean number of moderate/severe VMS episodes per 24 hours self-reported by participants via an an eDiary | Baseline to weeks 4, 8 and 12
  Participant manually records moderate/severe VMS episodes on the eDiary.
Mean change from baseline in the mean number of daytime moderate/severe VMS episodes per 24 hours self-reported by participants via an eDiary | Baseline to weeks 4, 8 and 12
  Participant manually records moderate/severe VMS episodes on the eDiary
Mean change from baseline in the mean number of nighttime moderate/severe VMS episodes per 24 hours self-reported by participants via an eDiary | Baseline to weeks 4, 8 and 12
  Participant manually records moderate/severe VMS episodes on the eDiary.
Number of participants with Adverse Events (AEs) | Up to 52 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a study drug, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal (investigational) product.
Number of participants with Serious Adverse Events (SAEs) | Up to 52 weeks
  An AE is considered "serious" if, in the view of either the investigator or sponsor, it:
  Results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, is a congenital anomaly or birth defect of a child conceived during the exposure of one of the parents to the drug studied, requires inpatient hospitalization or leads to prolongation of hospitalization, is a medically important event or reaction.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 52 weeks
  Number of participants with potentially clinically significant vital sign values.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development, Inc.
Locations (48):
- United States (48):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Accel Research Sites-Cahaba Medical Care-OBGYN, Birmingham, Alabama
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Torrance Clinical Research Institute,Inc, Lomita, California
  - Dream Team Clinical Research, Pomona, California
  - Wake Research - Medical Center for Clinical Research WR-MCCR, LLC, San Diego, California
  - Millennium Clinical Trials LLC, Simi Valley, California
  - Bayview Research Group, LLC, Valley Village, California
  - University of Colorado Health - Anschutz Cancer Pavilion - Anschutz Medical Campus, Aurora, Colorado
  - Accel Research Sites, DeLand, Florida
  - Nextlevel Research Center, Doral, Florida
  - Multi-Specialty Research Associates, Inc. (WR-MSRA, LLC), Lake City, Florida
  - Altus Research, Lake Worth, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Dr. Jarrett's Wellness Center, Miami, Florida
  - Complete Health Research, Ormond Beach, Florida
  - Comprehensive Clinical Trials, Llc, West Palm Beach, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Alpha Clinical Research Georgia, Dunwoody, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Chicago Clinical Research Institute Inc., Chicago, Illinois
  - Investigators Research Group, Llc, Brownsburg, Indiana
  - Praetorian Pharmaceutical Research, Marrero, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Montana Medical Research, Inc., Missoula, Montana
  - Bosque Women's Care, Albuquerque, New Mexico
  - Upstate Clinical Research Associates, Williamsville, New York
  - Premier Gynecology & Wellness, Charlotte, North Carolina
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Unified Women's Clinical Research, Winston-Salem, North Carolina
  - HWC Women's Research Center, Englewood, Ohio
  - Tekton Research, Moore, Oklahoma
  - Clinical Research Of Philadelphia, Llc, Philadelphia, Pennsylvania
  - Reading Hospital / Tower Health, West Reading, Pennsylvania
  - Biocentric Health Research, West Columbia, South Carolina
  - Chattanooga Medical Research, Llc, Chattanooga, Tennessee
  - Signature Gyn Services, Fort Worth, Texas
  - UT Health Women's Research Center at Memorial City, Houston, Texas
  - TMC Life Research, Inc, Houston, Texas
  - Biopharma Informatic Research Center, Houston, Texas
  - Pioneer Research Solutions, Inc, Houston, Texas
  - ClinRx Research LLC, Plano, Texas
  - DCT - Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Granger Medical Clinic, Riverton, Utah
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.